CLINICAL TRIAL: NCT03662217
Title: Personalized Nutrition for Diabetes Type 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DayTwo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003577
Record Dates: First submitted 2018-09-02; First posted 2018-09-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Type 2
Keywords: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algorithm-based diet (Experimental): Subjects randomized to this arm will receive personally tailored dietary recommendations based on their predicted glycemic responses according to the study algorithm.
  Interventions: Other: Algorithm-based diet
- ADA- based diet (Other): Subjects randomized to this arm will receive nutritional recommendations according to the standard American dietary approach for treating diabetes
  Interventions: Other: ADA- based diet

INTERVENTIONS:
Other: Algorithm-based diet — Personalized nutrition plan based on an algorithm for predicting the personalized glucose response to food. The algorithm's predictions are based on many personal measurements, including blood tests, personal lifestyle and gut bacteria
  Arms: Algorithm-based diet
Other: ADA- based diet — The American standard of care dietary guidelines for diabetes.
  Arms: ADA- based diet

SUMMARY:
The study will investigate the effect of personalized diet on blood glucose control in individuals with diabetes as compared with ADA diet.

The primary objective is to test whether personalized diets based on DayTwo's algorithm can improve glycemic control and metabolic health compared to standard ADA acceptable dietary approach for diabetes at the end of a 3-month intervention period.

DETAILED DESCRIPTION:
The prevalence of diabetes type 2 estimated to 628 Million people in the world by 2045 and was announced by the International Diabetes Federation (IDF) as one of the biggest epidemics in the history. Complications of diabetics Type 2 can range from high blood sugar include heart disease, strokes, diabetic retinopathy which can result in blindness, kidney failure, and poor blood flow in the limbs which may lead to amputations. It is also linked to other manifestations, collectively termed the metabolic syndrome, including obesity, hypertension, non-alcoholic fatty liver disease, hypertriglyceridemia and cardiovascular disease .

As blood glucose levels are mainly affected by food consumption, the growing number of blood glucose abnormalities is likely attributable to nutrition. Indeed, dietary and lifestyle changes normalize blood glucose levels in 55% -80% of the cases. Therefore, maintaining normal blood glucose levels is critical for preventing diabetes and its metabolic complications.

Currently, there are no effective methods for predicting the postprandial glycemic response (PPGR) of people to food. The current practice of using the meal carbohydrate content is a poor predictor of the PPGR and has limited efficacy. The glycemic index (GI), which quantifies PPGR to consumption of a single tested food type, and the derived glycemic load have limited applicability in assessing the PPGR to real-life meals consisting of arbitrary food combinations and varying quantities, consumed at different times of the day, and at different proximity to physical activity and other meals. Indeed, studies examining the effect of diets with a low glycemic index on TIIDM risk, weight loss, and cardiovascular risk factors yielded mixed results . The limited success of GI measure is probably due to the fact that it is a general index, which does not take into consideration the large variation between individuals in their glycemic response to food. It can be concluded, therefore, that in order to control glycemic response of an individual, we should build a personally tailored diet which takes into account various factors.

Although genetic factors influence the levels of fasting blood glucose and glycemic response to food, these factors only explain approximately 10% of the variance in the population. Supporting this claim is the fact that the number of people with diabetes is increasing in recent years regardless of patients' genetic background. In contrast, environmental factors such as the composition of the intestinal bacteria and their metabolic activity may affect the glycemic response. The entire bacteria population in the digestive tract (microbiome) consist of ~1,000 species with a genetic repertoire of ~3 million different genes. The microbiome is directly affected by our diet and directly affect the body's response to food. This special relationship between the host and the intestinal flora is reflected by the composition of bacteria unique to type 2 diabetes and in the significant changes in the bacteria composition upon transition from a diet rich in fiber to a "Western" diet rich in simple sugars.

Recently, DayTwo developed a highly accurate algorithm for predicting the personalized glucose response to food for each person based on the PNP Study conducted by the Weizmann Institute. The algorithm's predictions are based on many personal measurements, including blood tests, personal lifestyle and gut bacteria. In a small-scale pilot study that was conducted by the Weizmann Institute using the algorithm, the researchers personally tailored dietary interventions to healthy and prediabetic people, which resulted in significantly improved PPGRs accompanied by consistent alterations to the gut microbiota. These findings led to hypothesize that tailoring personalized diets based on PPGRs predictions may achieve better outcomes in terms of controlling blood glucose levels and its metabolic consequences relative to the current standard nutritional therapy for diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Type 2 for at least 1 year (diagnosed by ADA criteria) and up to 20 years
* 7.5 <= HbA1C <= 9.5
* Stable dose of meds for 3 months
* Stable diet and lifestyle for 3 months
* Age -between 18 to 85
* BMI - between 25 to 35
* Capable of working with smartphone application
* At least 5 days of the food logging in screening week:

  * At least 60% reported Kcals out of the recommended daily consumption
  * At least 2 reported meals a day

Exclusion Criteria:

* Short-acting insulin treatment
* Bariatric surgery
* Antibiotics/antifungal treatment in the last 3 months
* Use of weight-loss medication for less than 6 months
* Use of GLP-1 and SGLT-2 for less than 6 months
* People under another diet regime that is different from the ADA recommended diet
* Pregnancy or 3 months after giving birth, fertility treatments
* Chronic disease (e.g. HIV, Cushing syndrome, CKD, acromegaly, active hyperthyroidism etc.)
* Cancer and anticancer treatment in the last 5 years
* Psychiatric disorders (that in the eyes of the investigator should exclude the participant)
* Life-threatening food allergy
* Have received DayTwo nutrition recommendations in the past
* have been continuously using CGM\FGM
* Any disorder, which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-28 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Mean change in HbA1C from the baseline level | 3 months intervention period
  HbA1C
Evaluation of the total daily time of plasma glucose levels | 3 months intervention period
  Time in Range ▪ CGM glucose levels are between 70 to 180 mg/dl

SECONDARY OUTCOMES:
Evaluation of the total daily time of plasma glucose levels | 3 months intervention period
  Total daily time of CGM glucose levels below 70 mg/dl (Hypoglycemia incidents)
Evaluation of the total daily time of plasma glucose levels | 3 months intervention period
  Time in Range ▪ CGM glucose levels are between 70 to 140 mg/dl
Mean change in ADRR from the baseline level | 3 months intervention period
  ADRR
Mean change in BGRI from the baseline level | 3 months intervention period
  BGRI
Mean change in LBGI from the baseline level | 3 months intervention period
  LBGI
Mean change in HBGI from the baseline level | 3 months intervention period
  HBGI
Mean change in MAGE from the baseline level | 3 months intervention period
  MAGE
Mean change in CV glucose % from the baseline level | 3 months intervention period
  CV glucose %
Mean change in Glucose from the baseline level | 3 months intervention period
  Mean glucose
Mean change in Standard deviation of glucose from the baseline level | 3 months intervention period
  Standard deviation of glucose
Mean change in CONGA from the baseline level | 3 months intervention period
  CONGA
Change in Weight from baseline | 3 months intervention period
  Weight
Change in HbA1C from the baseline level | 3 months intervention period
  Percentage of patients with HbA1C <8%
Change in HbA1C from the baseline level | 3 months intervention period
  Percentage of patients with HbA1C <7%
change in HbA1C from the baseline level | 3 months intervention period
  Percentage of patients with HbA1C <6.5%
Change in Lipid profile parameters | 3 months intervention period
  Lipid profile
Change in Liver function parameters | 3 months intervention period
  Liver function test
Change in Creatinine parameter | 3 months intervention period
  Creatinine
Change in Fructosamin parameter | 3 months intervention period
  Fructosamin

OTHER OUTCOMES:
Patients satisfaction evaluation using Satisfaction questionnaire | 3 months intervention period
  Patients fill out Satisfaction questionnaire
Patients Diet compliance evaluation | 3 months intervention period
  Diet Compliance measure using food logging application

CONTACTS AND LOCATIONS:
Overall Officials: Davidi Bachrach, Study Director — DayTwo COO
Locations (2):
- Israel (2):
  - The Edith Wolfson Medical Center, Holon
  - Diabetes Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418